CLINICAL TRIAL: NCT04916873
Title: Rehabilitation Status of Children With Cerebral Palsy and Anxiety of Their Caregivers During the Covid19 Pandemic
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Akpınar, Assoc Prof, Fatih Sultan Mehmet Training and Research Hospital
Other Study IDs: FSMEAH-KAEK 2020/56
Record Dates: First submitted 2021-06-03; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy; Covid19; Anxiety
Keywords: Anxiety; Cerebral Palsy; Covid19; Rehabilitation
MeSH Terms: conditions — Cerebral Palsy; COVID-19; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rehabilitation status of children with cerebral palsy (CP) and anxiety of their caregivers during the covid19 pandemic were explored. 206 caregivers who voluntarily accepted to participate were administered the State-Trait Anxiety Inventory and evaluated about the rehabilitation status of their children.The anxiety levels of all caregivers were found high and the rehabilitation programmes of the children were interrupted.

DETAILED DESCRIPTION:
Investigators aimed to explore the rehabilitation status of children with CP and anxiety of their caregivers during the covid19 pandemic. Caregivers of children with CP who were under follow up in the outpatient CP clinic were called up during pandemic period. 206 caregivers who voluntarily accepted to participate were administered the State-Trait Anxiety Inventory and evaluated about the rehabilitation status of their children. Demographic data, associated problems of children, Gross Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS) levels were recorded from their files. For the statistical analysis, IBM SPSS Statistics 22 (SPSS IBM, Turkey) programs were used. While evaluating the study data, the suitability of the parameters to the normal distribution was evaluated with the Shapiro Wilks test. Significance was evaluated at the p <0.05 level.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children with CP who were under follow up in the outpatient CP clinic who voluntarily accepted to participate

Exclusion Criteria:

* Caregivers of children with CP who were under follow up in the outpatient CP clinic who didn't accept to participate

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Caregivers of children with CP who were under follow up in the outpatient CP clinic.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Anxiety of the caregivers of the children with cerebral palsy | 1 month
  State-Trait Anxiety levels of caregivers of the children with cerebral palsy during the covid19 pandemic.The total score of the State-Trait Anxiety scale varies between 20 and 80. Those who score below 36 are classified as "no anxiety", those between 37-42 points as "mild anxiety" and those with 42 points and above as "high anxiety".
Rehabilitation process of the children with cerebral palsy | 1 month
  Rehabilitation status of the children with cerebral palsy during the covid19 pandemic. Rehabilitation frequency of children and home exercise status are evaluated

CONTACTS AND LOCATIONS:
Overall Officials: PINAR AKPINAR, MD, Principal Investigator — Assoc Prof
Locations (1):
- Pinar Akpinar, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cacioppo M, Bouvier S, Bailly R, Houx L, Lempereur M, Mensah-Gourmel J, Kandalaft C, Varengue R, Chatelin A, Vagnoni J, Vuillerot C, Gautheron V, Dinomais M, Dheilly E, Brochard S, Pons C; ECHO Group. Emerging health challenges for children with physical disabilities and their parents during the COVID-19 pandemic: The ECHO French survey. Ann Phys Rehabil Med. 2021 May;64(3):101429. doi: 10.1016/j.rehab.2020.08.001. Epub 2020 Aug 18. PMID 32818674
- [Result] Dhiman S, Sahu PK, Reed WR, Ganesh GS, Goyal RK, Jain S. Impact of COVID-19 outbreak on mental health and perceived strain among caregivers tending children with special needs. Res Dev Disabil. 2020 Dec;107:103790. doi: 10.1016/j.ridd.2020.103790. Epub 2020 Oct 6. PMID 33091712